CLINICAL TRIAL: NCT02366143
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab (MPDL3280A, Anti-PD-L1 Antibody) in Combination With Carboplatin+Paclitaxel With or Without Bevacizumab Compared With Carboplatin + Paclitaxel + Bevacizumab in Chemotherapy-Naïve Patients With Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in Combination With Carboplatin Plus (+) Paclitaxel With or Without Bevacizumab Compared With Carboplatin+Paclitaxel+Bevacizumab in Participants With Stage IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Acronym: IMpower150
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29436; 2014-003207-30 (EudraCT Number)
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Bevacizumab; Carboplatin; Paclitaxel

ARMS (3):
- Arm A (Atezolizumab+Paclitaxel+Carboplatin) (Experimental): Participants received intravenous (IV) infusion of atezolizumab on Day 1 of each 21-day cycle followed by IV infusion of paclitaxel and carboplatin on Day 1 of each 21-day cycle for 4 or 6 cycles or until loss of clinical benefit whichever occurs first, during induction treatment phase. Participants received IV infusion of atezolizumab during maintenance treatment phase until loss of clinical benefit.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) (Experimental): Participants received IV infusion of atezolizumab and bevacizumab on Day 1 of each 21-day cycle followed by IV infusion of paclitaxel and carboplatin on Day 1 of each 21-day cycle for 4 or 6 cycles or until loss of clinical benefit whichever occurs first, during induction treatment phase. Participants received IV infusion of atezolizumab until loss of clinical benefit and bevacizumab until progressive disease, unacceptable toxicity, or death during maintenance treatment phase.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- Arm C (Bevacizumab+Paclitaxel+Carboplatin) (Active Comparator): Participants received IV infusion of bevacizumab on Day 1 of each 21-day cycle followed by IV infusion of paclitaxel and carboplatin on Day 1 of each 21-day cycle for 4 or 6 cycles or loss of clinical benefit whichever occurs first, during induction treatment phase. Participants received IV infusion of bevacizumab during maintenance treatment phase until progressive disease, unacceptable toxicity, or death.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab was administered as IV infusion at a dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle until loss of clinical benefit.
  Other Names: MPDL3280A; RO5541267; Tecentriq
  Arms: Arm A (Atezolizumab+Paclitaxel+Carboplatin); Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin)
Drug: Bevacizumab — Bevacizumab was administered as IV infusion at a dose of 15 milligrams per kilogram (mg/kg) on Day 1 of each 21-day cycle until progressive disease, unacceptable toxicity, or death.
  Arms: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin); Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Drug: Carboplatin — Carboplatin was administered at area under the concentration-time curve (AUC) 6 milligrams per milliliter per minute (mg/mL/min) on Day 1 of each 21-day cycle for 4 or 6 cycles or until loss of clinical benefit whichever occurs first.
Drug: Paclitaxel — Paclitaxel was administered as IV infusion at a dose of 200 milligrams per square meter (mg/m^2) on Day 1 of each 21-day cycle for 4 or 6 cycles or until loss of clinical benefit whichever occurs first.

SUMMARY:
This randomized, open-label study evaluated the safety and efficacy of atezolizumab (an engineered anti-programmed death-ligand 1 [PD-L1] antibody) in combination with carboplatin+paclitaxel with or without bevacizumab compared with treatment with carboplatin+paclitaxel+bevacizumab in chemotherapy-naïve participants with Stage IV non-squamous NSCLC. Participants were randomized in a 1:1:1 ratio to Arm A (Atezolizumab+Carboplatin+Paclitaxel), Arm B (Atezolizumab+Carboplatin+Paclitaxel+Bevacizumab), or Arm C (Carboplatin+Paclitaxel+Bevacizumab).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status 0 or 1
* Histologically or cytologically confirmed, Stage IV non-squamous NSCLC
* Participants with no prior treatment for Stage IV non-squamous NSCLC
* Known PD-L1 status as determined by immunohistochemistry assay performed on previously obtained archival tumor tissue or tissue obtained from a biopsy at screening
* Measurable disease as defined by RECIST v1.1
* Adequate hematologic and end organ function

Exclusion Criteria:

Cancer-Specific Exclusions:

* Active or untreated central nervous system metastases
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome

General Medical Exclusions:

* Pregnant or lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Severe infection within 4 weeks prior to randomization
* Significant cardiovascular disease
* Illness or condition that interferes with the participant's capacity to understand, follow and/or comply with study procedures

Exclusion Criteria Related to Medications:

* Prior treatment with cluster of differentiation 137 agonists or immune checkpoint blockade therapies, anti-programmed death-1, and anti-PD-L1 therapeutic antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (240):
- United States (61):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Arizona Oncology Associates, Flagstaff, Arizona
  - Southern CA Permanente Med Grp, Bellflower, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Scripps Health, La Jolla, California
  - Chao Family Comprehensive Cancer Center UCI, Orange, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Kaiser Permanente, Lonetree, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Holy Cross Hospital Inc, Fort Lauderdale, Florida
  - Cancer Specialists of North Florida - Baptist South, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Univ of Chicago, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Hematology-Oncology; Associates of the Quad Cities, Bettendorf, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - New England Cancer Specialists, Scarborough, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Regional Cancer Care Associates, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - St. Joseph Mercy Health System, Ann Arbor, Michigan
  - St. Luke's Regional Cancer Center, Duluth, Minnesota
  - Park Nicolett - Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Valley Hospital; Oncology Research, Paramus, New Jersey
  - Regional Cancer Care Associates LLC, Sewell, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - First Health of the Carolinas, Pinehurst, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Mercy St Anne Hospital, Toledo, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - St. Charles Medical Center Bend; Cancer Care Of The Cascades, Bend, Oregon
  - Willamette Valley Cancer Insitute and Research Center, Springfield, Oregon
  - St. Luke's Cancer Care Associates, Bethlehem, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Medical Ctr, Pittsburgh, Pennsylvania
  - West Clinic, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
  - West Virginia University; Mary Babb Randolph Can Ctr, Morgantown, West Virginia
- Argentina (7):
  - Centro Medico Austral, Buenos Aires
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Sanatorio Allende, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Hospital Provincial del Centenario, Rosario
  - Fundacion Koriza, Santa Rosa
  - Centro de Investigacion; Clinica - Clinica Viedma S.A., Viedma
- Australia (16):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Cancer Care Centre, Sydney, New South Wales
  - Prince Charles Hospital; Department of Medical Oncology, Chermside, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Frankston Hospital, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - The Alfred Hospital, Prahan, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (2):
  - Paracelsus Medizinische Privatuniversität, Salzburg
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (2):
  - CHU de Liège, Liège
  - Clinique Ste-Elisabeth, Namur
- Brazil (9):
  - CETUS Hospital Dia Oncologia, Uberaba, Minas Gerais
  - Instituto Do Cancer Delondrina_X; Unidade De Pesquisa Clinica, Londrina, Paraná
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - IPCEM; Instituto de Pesquisa de Estudos Multicêntricos, Caxias do Sul, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto Ribeirãopretano de Combate Ao Câncer; Centro Especializado De Oncologia, Ribeirão Preto, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital A. C. Camargo; Oncologia, São Paulo, São Paulo
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - MHAT Serdika, EOOD, Sofia
- Lakeridge Health Center, Oshawa, Ontario, Canada
- Chile (3):
  - Clinica Santa Maria, Santiago
  - Health & Care SPA, Santiago
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
- France (12):
  - Institut Bergonié Centre Régional de Lutte Contre Le Cancer de Bordeaux Et Sud Ouest, Bordeaux
  - CHU de Grenoble, Grenoble
  - Centre Jean Bernard Clinique Victor Hugo, Le Mans
  - Hôpital Saint Joseph, Marseille
  - Hopital Nord AP-HM, Marseille
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Bordeaux, Pessac
  - Service de Pneumologie Centre Hospitalier Régional La Réunion Site Felix Guyon, Saint-Denis
  - CH de Saint Quentin, Saint-Quentin
  - Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer, Toulon
  - Hôpital d'Instruction des Armées de Sainte Anne; Service de Pneumologie, Toulon
  - Hôpital Larrey;Université Paul Sabatier, Toulouse
- Germany (17):
  - Zentralklinikum Augsburg, Augsburg
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Ev.Krankenhaus Bielefeld gGmbH; Klinik für Innere Medizin und Geriatrie, Bielefeld
  - Augusta Kranken-Anstalt gGmbH, Bochum
  - Kliniken der Stadt Koln gGmbH; Lungenklinik Onkologische Ambulanz, Cologne
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - St. Elisabethen Krankenhaus, Frankfurt am Main
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria; Halle-Dolau gGmbH, Halle
  - Asklepios Klinik Harburg, Hamburg
  - Lungenklinik Hemer, Hemer
  - Universität Des Saarlandes; Klinik für Innere Medizin V, Homburg
  - Klinik Loewenstein gGmbH; Onk & Pal, Löwenstein
  - Klinikum Bogenhausen, München
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
  - Klinikum der Universität Regensburg, Regensburg
  - Stiftung Mathias-Spital Rheine, Rheine
- Italy (11):
  - AORN A Cardarelli, Napoli, Campania
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Università Cattolica Del S Cuore, Rome, Lazio
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genoa, Liguria
  - ASL 3 Genovese; DSM, Genoa, Liguria
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Unita Sanitaria Locale N1 Sassari; Unita Operativa Di Oncologia Medica, Sassari, Sardinia
  - Policlinico Vittorio Emanuele, Catania, Sicily
  - Ospedale Versilia, Lido di Camaiore, Tuscany
  - Ospedale Civile - Livorno, Livorno, Tuscany
- Japan (15):
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - NHO Kyushu Cancer Center, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Miyagi Cancer Center, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka City University Hospital, Osaka
  - National Hospital Organization Osaka Toneyama Medical Center, Osaka
  - Toranomon Hospital, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Kyorin University Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital Latvian Oncology Centre, Riga
- National Cancer Institute, Vilnius, Lithuania
- Mexico (3):
  - Centro Universitario Contra El Cancer, Monterrey
  - Cancerologia de Queretaro, Querétaro
  - Centro Hemato Oncologico Privado; Oncologia, Toluca
- Netherlands (12):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Amsterdam UMC Location VUMC, Amsterdam
  - Amphia Ziekenhuis; Afdeling Longziekten, Breda
  - Ziekenhuis Gelderse Vallei, Ede
  - Tergooiziekenhuizen, Hilversum
  - Spaarne Gasthuis; Spaarne Ziekenhuis, Hoofddorp
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Ziekenhuis; R&D Long, Nieuwegein
  - Erasmus MC; Afdeling Longziekten, Rotterdam
  - Maasstad ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Gelre Ziekenhuizen, Zutphen, Zutphen
- Peru (3):
  - Centro Medico Monte Carmelo, Arequipa
  - Centro Especializado de Enfermedades Neoplásicas, Arequipa
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
- Portugal (6):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Instituto Portugues Oncologia de Lisboa Francisco Gentil EPE, Lisbon
  - Hospital Pulido Valente; Servico de Pneumologia, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
  - Hospital de Sao Joao; Servico de Pneumologia, Porto
- Russia (5):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Russian Oncology Research Center n.a. N.N. Blokhin, Moscow
  - Clinical Oncology Dispensary, Omsk
  - Evromedservis LCC, Pushkin
  - City Clinical Oncology Dispensary, Saint Petersburg
- National Cancer Centre; Medical Oncology, Singapore, Singapore
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Narodny onkologicky ustav, Bratislava
  - POKO Poprad s.r.o., Poprad
- Spain (20):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Instituto Catalan de Oncologia de Hospitalet (ICO); Servicio de Farmacia, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, LAS Palmas
  - Complejo Hospitalario U. de Ourense, Ourense, Orense
  - Hospital Lluis Alcanyis De Xativa, Xàtiva, Valencia
  - Hospital del Mar, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Lucus Augusti; Servicio de Oncologia, Lugo
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario Fundación Jimenez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (3):
  - Kantonsspital Baselland, Bruderholz
  - Luzerner Kantonsspital Sursee, Lucerne
  - Kantonsspital St. Gallen; Onkologie/Hämatologie, Sankt Gallen
- Taiwan (10):
  - Changhua Christian Hospital; Hematology-Oncology, Changhua
  - Kaohsiung Medical University Hospital; Department of Urology, Kaohsiung City
  - Chi Mei Medical Center Liou Ying Campus, Liuying Township
  - Chang Gung Memorial Hospital Chiayi, Putzu
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan Uni Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
  - Taichung Veterans General Hospital, Xitun Dist.
- Ukraine (13):
  - ME Bukovinian Clinical Oncology Center, Chernivtsi, Chernihiv Governorate
  - Municipal Institution City Clinical Hospital #4 of Dnipro City Council - PPDS; Dept of Chemotherapy, Dnipropetrovsk, Katerynoslav Governorate
  - Uzhgorod Central City Clinical Hospital, Uzhhorod, Katerynoslav Governorate
  - MNPE Zaporizhzhia Regional Antitumor Center ZRC, Zaporizhzhia, Katerynoslav Governorate
  - Communal Non profit Enterprise Regional Center of Oncology; Oncosurgical dept of thoracic organs, Kharkiv, Kharkiv Governorate
  - MNPE Transcarpathian Antitumor Center of the Transcarpathian Regional Council; Chemotherapy Dept, Uzhhorod, Kherson Governorate
  - Municipal Institution SubCarpathian Clinical Oncological Centre; Surgical department#2, Ivano-Frankivsk, KIEV Governorate
  - Communal Nonprofit Enterprise Podilsky Regional Center Of Oncology OfTheVinnytsia Regional Council, Vinnytsia, KIEV Governorate
  - SI Institute of Medical Radiology n.a. S.P. Hryhoriev of NAMS of Ukraine, Kharkiv
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs'k Regional Council; Chemotherapy Department, Kryvyi Rih
  - Kyiv City Clinical Oncological Center, Kyiv
  - Poltava Regional Clinical Oncology Dispensary of Poltava Regional Council; Thoracic department, Poltava
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy

REFERENCES:
- [Derived] Zhou C, Dong X, Chen G, Wang Z, Wu X, Yao Y, Zhang Y, Cheng Y, Pan H, Zhang X, Cui J, Wang L, Chen X, Li X, Wang Z, Wang Q, He J, Wang M, Yan I, Qian L, Xu M, Huang X, Sun C, Cai J, Wu Q, Ballinger M, Kaul M, Srivastava MK. Atezolizumab plus bevacizumab and chemotherapy in metastatic nonsquamous NSCLC: the randomized double-blind phase 3 IMpower151 trial. Nat Med. 2025 Jul;31(7):2375-2384. doi: 10.1038/s41591-025-03658-y. Epub 2025 May 16. PMID 40379995
- [Derived] Mang A, Zou W, Rolny V, Reck M, Cigoianu D, Schulze K, Holdenrieder S, Socinski MA, Shames DS, Wehnl B, Patil NS. Combined use of CYFRA 21-1 and CA 125 predicts survival of patients with metastatic NSCLC and stable disease in IMpower150. Tumour Biol. 2024;46(s1):S177-S190. doi: 10.3233/TUB-230001. PMID 37545290
- [Derived] Socinski MA, Jotte RM, Cappuzzo F, Nishio M, Mok TSK, Reck M, Finley GG, Kaul MD, Yu W, Paranthaman N, Bara I, West HJ. Association of Immune-Related Adverse Events With Efficacy of Atezolizumab in Patients With Non-Small Cell Lung Cancer: Pooled Analyses of the Phase 3 IMpower130, IMpower132, and IMpower150 Randomized Clinical Trials. JAMA Oncol. 2023 Apr 1;9(4):527-535. doi: 10.1001/jamaoncol.2022.7711. PMID 36795388
- [Derived] Ton TGN, Pal N, Trinh H, Mahrus S, Bretscher MT, Machado RJM, Sadetsky N, Chaudhary N, Lu MW, Riely GJ. Replication of Overall Survival, Progression-Free Survival, and Overall Response in Chemotherapy Arms of Non-Small Cell Lung Cancer Trials Using Real-World Data. Clin Cancer Res. 2022 Jul 1;28(13):2844-2853. doi: 10.1158/1078-0432.CCR-22-0471. PMID 35511917
- [Derived] Nogami N, Barlesi F, Socinski MA, Reck M, Thomas CA, Cappuzzo F, Mok TSK, Finley G, Aerts JG, Orlandi F, Moro-Sibilot D, Jotte RM, Stroyakovskiy D, Villaruz LC, Rodriguez-Abreu D, Wan-Teck Lim D, Merritt D, Coleman S, Lee A, Shankar G, Yu W, Bara I, Nishio M. IMpower150 Final Exploratory Analyses for Atezolizumab Plus Bevacizumab and Chemotherapy in Key NSCLC Patient Subgroups With EGFR Mutations or Metastases in the Liver or Brain. J Thorac Oncol. 2022 Feb;17(2):309-323. doi: 10.1016/j.jtho.2021.09.014. Epub 2021 Oct 7. PMID 34626838
- [Derived] Socinski MA, Nishio M, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kong S, Lee A, Coleman S, Zou W, McCleland M, Shankar G, Reck M. IMpower150 Final Overall Survival Analyses for Atezolizumab Plus Bevacizumab and Chemotherapy in First-Line Metastatic Nonsquamous NSCLC. J Thorac Oncol. 2021 Nov;16(11):1909-1924. doi: 10.1016/j.jtho.2021.07.009. Epub 2021 Jul 24. PMID 34311108
- [Derived] Reck M, Wehler T, Orlandi F, Nogami N, Barone C, Moro-Sibilot D, Shtivelband M, Gonzalez Larriba JL, Rothenstein J, Fruh M, Yu W, Deng Y, Coleman S, Shankar G, Patel H, Kelsch C, Lee A, Piault E, Socinski MA. Safety and Patient-Reported Outcomes of Atezolizumab Plus Chemotherapy With or Without Bevacizumab Versus Bevacizumab Plus Chemotherapy in Non-Small-Cell Lung Cancer. J Clin Oncol. 2020 Aug 1;38(22):2530-2542. doi: 10.1200/JCO.19.03158. Epub 2020 May 27. PMID 32459597
- [Derived] Reck M, Mok TSK, Nishio M, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Lee A, Coleman S, Deng Y, Kowanetz M, Shankar G, Lin W, Socinski MA; IMpower150 Study Group. Atezolizumab plus bevacizumab and chemotherapy in non-small-cell lung cancer (IMpower150): key subgroup analyses of patients with EGFR mutations or baseline liver metastases in a randomised, open-label phase 3 trial. Lancet Respir Med. 2019 May;7(5):387-401. doi: 10.1016/S2213-2600(19)30084-0. Epub 2019 Mar 25. PMID 30922878
- [Derived] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm C: Bevacizumab+Paclitaxel+Carboplatin
- Arm B: Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin
- Arm A: Atezolizumab+Paclitaxel+Carboplatin
Period: Overall Study
Arm/Group | Arm C | Arm B | Arm A
Started | 400 | 400 | 402
Completed | 0 | 0 | 0
Not Completed | 400 | 400 | 402
Not completed — Death | 307 | 278 | 280
Not completed — Lost to Follow-up | 2 | 4 | 2
Not completed — Physician Decision | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 16 | 17 | 22
Not completed — Sponsor request to withdraw/discontinue patient | 0 | 6 | 0
Not completed — Increased Microscopic RBCS on Urinalysis | 0 | 1 | 0
Not completed — Randomization Error | 1 | 0 | 0
Not completed — PI Move and Site Closure | 1 | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 0 | 2
Not completed — Sponsor request to withdraw/discontinue patient in survival follow up | 70 | 57 | 52
Not completed — Patient moved to roll-over study | 1 | 19 | 28
Not completed — Patient moved to commercial stock | 0 | 0 | 1
Not completed — Patient stopped treatment due to disease progression;didn't enter follow up due to study termination | 0 | 0 | 1
Not completed — Patient rolling over to patient assistance program | 0 | 0 | 1
Not completed — Patient continue same treatment via Post Trial Access Progarm (PTAP) | 0 | 0 | 1
Not completed — Requester's instructions | 1 | 1 | 1
Not completed — Uneligible | 0 | 1 | 0
Not completed — Post Trial Migration | 0 | 1 | 0
Not completed — Patient moving onto PTAP commercial stock | 0 | 1 | 0
Not completed — Patient switched to PTAP | 0 | 1 | 0
Not completed — Patient moved to commercial atezolizumab use | 0 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm C | Arm B | Arm A | Total
Number analyzed (Participants) | 400 | 400 | 402 | 1202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (9.3) | 63.0 (9.5) | 62.3 (9.2) | 62.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 160 | 161 | 482
  Male | 239 | 240 | 241 | 720
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 46 | 56 | 48 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 3 | 9 | 24
  White | 335 | 322 | 331 | 988
  More than one race | 0 | 3 | 4 | 7
  Unknown or Not Reported | 6 | 13 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS), as Determined by the Investigator in Arm B Versus Arm C in the Teff-high WT Population and ITT-WT Population
Description: Progression Free Survival (PFS), as Determined by the Investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Arm B versus Arm C in the T-effector (Teff)-high wild type (WT) population and the intent-to-treat (ITT)-WT population.
Time Frame: Baseline until disease progression or death, whichever occurs first until data cut-off on 15 September 2017 (up to approximately 29 months)
Population: Teff-high WT population is defined as the Teff-high population excluding patients with an activating EGFR mutation or ALK translocation. ITT-WT population is defined as the ITT population excluding patients with an activating EGFR mutation or ALK translocation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 356 | 336
Months
  Teff-high WT Population: number analyzed (Participants) | 155 | 129
  Teff-high WT Population | 11.3 [9.1 to 13.0] | 6.8 [5.9 to 7.4]
  ITT-WT Population | 8.3 [7.7 to 9.8] | 6.8 [6.0 to 7.1]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT-WT population; Test type: Superiority — Stratified Analysis; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.52 to 0.74]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff-high WT Population; Test type: Superiority — Stratified Analysis; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.38 to 0.68]

2. Primary Outcome: Overall Survival (OS) in Arm B Versus Arm C in ITT-WT Population
Description: Overall Survival (OS) in Arm B Versus Arm C in ITT-WT Population
Time Frame: Baseline until death until data cut-off on 22 January 2018 (up to approximately 34 months)
Population: ITT-WT population is defined as the ITT population excluding patients with an activating EGFR mutation or ALK translocation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 359 | 337
Months | 19.2 [17.0 to 23.8] | 14.7 [13.3 to 16.9]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p = 0.0164, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.64 to 0.96]

3. Primary Outcome: Overall Survival (OS) in Arm A Versus Arm C in ITT-WT Population
Description: Overall Survival (OS) in Arm A Versus Arm C in ITT-WT Population
Time Frame: Baseline until death (up approximately 53 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 350 | 338
Months | 19.0 [15.7 to 21.5] | 14.7 [12.9 to 17.1]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p = 0.0528, Log Rank; Hazard Ratio (HR) = 0.842, 95% CI 2-sided [0.707 to 1.002]

4. Secondary Outcome: PFS, as Determined by the Independent Review Facility (IRF) in Arm B Versus Arm C in Teff-High-WT Population and ITT-WT Population
Description: PFS, as determined by the independent review facility (IRF) Using RECIST v1.1 in Arm B versus Arm C in the T-effector (Teff)-high wild type (WT) population and the intent-to-treat (ITT)-WT population.
Time Frame: Baseline until disease progression or death, whichever occurs first (up to approximately 29 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 356 | 336
Months
  Teff-high WT Population: number analyzed (Participants) | 155 | 129
  Teff-high WT Population | 10.7 [8.4 to 13.0] | 7.0 [6.1 to 8.1]
  ITT-WT Population | 8.5 [7.7 to 9.7] | 7.0 [6.3 to 8.0]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT-WT population; Test type: Superiority — Stratified Analysis; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.59 to 0.85]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.564, 95% CI 2-sided [0.418 to 0.760]

5. Secondary Outcome: PFS, as Determined by the Investigator in Arm B Versus Arm C in Teff High Population and ITT Population
Description: PFS, as determined by the investigator according to RECIST v1.1, in Arm B versus C in the Teff high population and ITT population.
Time Frame: Baseline until disease progression or death, whichever occurs first (up to approximately 29 months)
Population: Teff-high population is defined as the patients in the ITT population with Teff signature expression >=-1.91. ITT population is defined as all randomized patients, regardless of receipt of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 400 | 400
Months
  Teff-high Population: number analyzed (Participants) | 166 | 148
  Teff-high Population | 11.3 [9.1 to 13.0] | 6.8 [5.8 to 7.3]
  ITT Population | 8.3 [7.9 to 9.8] | 6.8 [6.0 to 7.1]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff-high Population; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.492, 95% CI 2-sided [0.374 to 0.649]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT Population; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.610, 95% CI 2-sided [0.517 to 0.720]

6. Secondary Outcome: PFS, as Determined by the Investigator in Arm A Versus Arm B in Teff High-WT Population and ITT-WT Population
Description: PFS, as determined by the investigator according to RECIST v1.1, in Arm A versus B in the Teff high-WT population and ITT-WT population.
Time Frame: Baseline until disease progression or death, whichever occurs first (up to approximately 29 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin)
Number analyzed (Participants) | 348 | 356
Months
  Teff-high WT: number analyzed (Participants) | 161 | 155
  Teff-high WT | 6.3 [5.6 to 7.8] | 11.3 [9.1 to 13.0]
  ITT-WT | 6.3 [5.6 to 7.0] | 8.3 [7.7 to 9.8]

7. Secondary Outcome: PFS, as Determined by the Investigator in Arm B Versus Arm C by PD-L1 Subgroup
Description: PFS as Determined by the Investigator according to RECIST v1.1, in Arm B Versus Arm C by PD-L1 Subgroup: TC2/3 or 1C2/3 and TC1/2/3 or IC1/2/3 (ITT-WT Population)
Time Frame: Baseline until disease progression or death, whichever occurs first (up to approximately 29 months)
Population: The PD-L1-selected WT populations are defined as the PD-L1-selected populations (TC2/3 or IC2/3 population or TC1/2/3 or IC1/2/3 population) excluding patients with a sensitizing EGFR mutation or ALK translocation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 190 | 164
Months
  TC2/3 or IC2/3 Subgroup: number analyzed (Participants) | 129 | 115
  TC2/3 or IC2/3 Subgroup | 11.1 [8.3 to 13.0] | 6.8 [5.8 to 7.7]
  TC1/2/3 or IC1/2/3 Subgroup | 11.0 [8.3 to 12.5] | 6.8 [5.8 to 7.3]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); TC2/3 or IC2/3 Subgroup; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.471, 95% CI 2-sided [0.352 to 0.647]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 Subgroup; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.486, 95% CI 2-sided [0.386 to 0.639]

8. Secondary Outcome: OS in Arm B Versus Arm C by PD-L1 Subgroup
Description: OS in Arm B Versus Arm C by PD-L1 Subgroup: TC2/3 or 1C2/3 and TC1/2/3 or IC1/2/3 (ITT-WT Population)
Time Frame: Baseline until death (up to approximately 34 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 192 | 165
Months
  TC 2/3 or IC2/3 Population: number analyzed (Participants) | 129 | 116
  TC 2/3 or IC2/3 Population | 22.2 [17.0 to 26.1] | 16.7 [10.5 to 24.2]
  TC1/2/3 or IC1/2/3 Population | 22.5 [18.2 to 26.1] | 16.4 [11.2 to 22.9]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); TC2/3 or IC2/3, WT ITT; Test type: Superiority — Unstratified Analysis; p = 0.2765, Log Rank; Hazard Ratio (HR) = 0.824, 95% CI 2-sided [0.580 to 1.169]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3, WT ITT; Test type: Superiority — Unstratified Analysis; p = 0.0829, Log Rank; Hazard Ratio (HR) = 0.771, 95% CI 2-sided [0.575 to 1.035]

9. Secondary Outcome: OS in Arm A Versus Arm C by PD-L1 Subgroup
Description: OS in Arm A Versus Arm C by PD-L1 Subgroup: TC2/3 or 1C2/3 and TC1/2/3 or IC1/2/3 (ITT-WT Population)
Time Frame: Baseline until death (up approximately 53 months)
Population: PD-L1 WT populations are defined as the PD-L1 populations (TC2/3 or IC2/3 population or TC1/2/3 or IC1/2/3 population) excluding patients with an activating EGFR mutation or ALK translocation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 185 | 165
Months
  TC2/3 or IC2/3 Population: number analyzed (Participants) | 124 | 116
  TC2/3 or IC2/3 Population | 26.1 [20.5 to 40.0] | 17.0 [10.3 to 22.9]
  TC1/2/3 or IC1/2/3 Population | 24.4 [20.2 to 28.1] | 16.0 [11.2 to 20.1]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT-WT; Test type: Superiority — Unstratified Analysis; p = 0.0073, Log Rank; Hazard Ratio (HR) = 0.709, 95% CI 2-sided [0.551 to 0.913]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); TC2/3 or IC2/3 Population; Test type: Superiority — Unstratified Analysis; p = 0.0097, Log Rank; Hazard Ratio (HR) = 0.662, 95% CI 2-sided [0.484 to 0.907]

10. Secondary Outcome: OS in Arm B Versus Arm C in Teff High-WT Population, Teff High Population, and ITT Population
Time Frame: Baseline until death (up to approximately 34 months)
Population: Teff-high WT population, defined as the Teff-high population excluding patients with activating EGFR mutation or ALK translocation. Teff-high population, defined as participants in the ITT population with Teff signature expression >=-1.91. ITT population, defined as all randomized patients, regardless of receipt of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 400 | 400
Months
  Teff High-WT Population: number analyzed (Participants) | 156 | 129
  Teff High-WT Population | 25.0 [17.8 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 16.7 [12.4 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Teff High Population: number analyzed (Participants) | 166 | 148
  Teff High Population | 25.2 [19.1 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 16.7 [12.4 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  ITT Population | 19.8 [17.4 to 24.2] | 14.9 [13.4 to 17.1]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff high-WT; Test type: Superiority — Stratified Analysis; p = 0.2843, Log Rank; Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.592 to 1.167]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff high; Test type: Superiority — Stratified Analysis; p = 0.1861, Log Rank; Hazard Ratio (HR) = 0.802, 95% CI 2-sided [0.579 to 1.113]
Statistical Analysis 3: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT; Test type: Superiority — Stratified Analysis; p = 0.0060, Log Rank; Hazard Ratio (HR) = 0.764, 95% CI 2-sided [0.630 to 0.926]

11. Secondary Outcome: OS in Arm A Versus Arm C in Teff High-WT Population, Teff High Population, and ITT Population
Time Frame: Baseline until death (up approximately 53 months)
Population: Teff-high WT population, defined as Teff-high population excluding patients with an activating EGFR mutation or ALK translocation. Teff-high population, defined as patients in the ITT population with Teff signature expression >=-1.91. ITT population is defined as all randomized patients, regardless of receipt of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 402 | 400
Months
  Teff-high WT Population: number analyzed (Participants) | 163 | 130
  Teff-high WT Population | 21.3 [17.6 to 26.3] | 16.3 [11.2 to 22.3]
  Teff-high Population: number analyzed (Participants) | 177 | 148
  Teff-high Population | 21.0 [17.1 to 26.0] | 16.7 [11.4 to 21.6]
  ITT Population | 19.0 [16.3 to 21.5] | 15.0 [13.4 to 17.1]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff high-WT; Test type: Superiority — Stratified Analysis; p = 0.0894, Log Rank; Hazard Ratio (HR) = 0.786, 95% CI 2-sided [0.595 to 1.038]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff high; Test type: Superiority — Stratified Analysis; p = 0.1276, Log Rank; Hazard Ratio (HR) = 0.815, 95% CI 2-sided [0.626 to 1.061]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT; Test type: Superiority — Stratified Analysis; p = 0.0681, Log Rank; Hazard Ratio (HR) = 0.861, 95% CI 2-sided [0.733 to 1.011]

12. Secondary Outcome: OS in Arm A Versus Arm B in Teff High-WT Population and ITT-WT Population
Time Frame: Baseline until death (up approximately 53 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin)
Number analyzed (Participants) | 350 | 359
Months
  Teff High-WT Population: number analyzed (Participants) | 163 | 156
  Teff High-WT Population | 21.3 [17.6 to 26.3] | 25.8 [19.1 to 32.6]
  ITT-WT Population | 19.0 [15.7 to 21.5] | 19.5 [17.0 to 22.2]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin); Teff high-WT ITT; Test type: Superiority — Stratified Analysis; p = 0.4599, Log Rank; Hazard Ratio (HR) = 0.901, 95% CI 2-sided [0.683 to 1.188]

13. Secondary Outcome: Duration of Response (DOR), as Determined By Investigator in Arm B Versus Arm C
Description: DOR, as determined by investigator according to RECIST v1.1 in Arm B versus Arm C in the Teff high-WT population and the ITT-WT population.
Time Frame: Baseline until disease progression or death, whichever occurs first (up to approximately 29 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 224 | 159
Months
  Teff high-WT Population: number analyzed (Participants) | 106 | 68
  Teff high-WT Population | 11.2 [9.7 to 15.7] | 5.7 [4.9 to 7.0]
  ITT-WT Population | 9.0 [6.9 to 11.4] | 5.7 [5.1 to 6.5]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT-WT; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.523, 95% CI 2-sided [0.406 to 0.675]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff-high WT; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.420, 95% CI 2-sided [0.283 to 0.624]

14. Secondary Outcome: Percentage of Participants With an Objective Response (OR) (Complete Response [CR] or Partial Response [PR]) as Determined by the Investigator in the Teff-High-WT Population and ITT-WT Population
Description: Percentage of Participants With an Objective Response (OR) (Complete Response [CR] or Partial Response [PR]) as Determined by the Investigator using RECIST v1.1 in the Teff-High-WT population and ITT-WT population.
Time Frame: Baseline until disease progression or death, whichever occurs first (up to approximately 29 months)
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 347 | 353 | 331
Percentage
  Teff-high WT Population: number analyzed (Participants) | 161 | 153 | 127
  Teff-high WT Population | 54.0 | 69.3 | 53.5
  ITT-WT Population | 49.3 | 63.5 | 48.0

15. Secondary Outcome: OS Rates at Years 1 and 2 in Arm B Versus Arm C
Description: OS at 1- and 2-year landmark timepoints in Teff-high WT population and ITT-WT population.
Time Frame: Baseline to 2 years or death, whichever occurs first.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 235 | 196
Percentage
  1-Year Teff-high WT Population: number analyzed (Participants) | 105 | 71
  1-Year Teff-high WT Population | 68.63 [61.28 to 75.98] | 58.74 [50.03 to 67.45]
  1-Year ITT-WT Population | 67.32 [62.41 to 72.22] | 60.63 [55.34 to 65.93]
  2-Year Teff-high WT Population: number analyzed (Participants) | 21 | 15
  2-Year Teff-high WT Population | 52.03 [43.12 to 60.94] | 41.70 [31.55 to 51.85]
  2-Year ITT-WT Population: number analyzed (Participants) | 34 | 29
  2-Year ITT-WT Population | 43.42 [36.94 to 49.90] | 33.71 [27.44 to 39.98]
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 1-Year ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.0697, Z-test; Difference in Event Free Rate = 6.68, 95% CI 2-sided [-0.54 to 13.90]
Statistical Analysis 2: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 2-Year ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.0347, Z-test; Difference in Event Free Rate = 9.71, 95% CI 2-sided [0.70 to 18.73]
Statistical Analysis 3: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 1-Year Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.0890, Z-test; Difference in Event Free Rate = 9.89, 95% CI 2-sided [-1.51 to 21.29]
Statistical Analysis 4: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 2-Year Teff-high WT Population; Test type: Other — Stratified Analysis; p = 0.1336, Z-test; Difference in Event Free Rate = 10.34, 95% CI 2-sided [-3.17 to 23.84]

16. Secondary Outcome: OS Rates at Years 1 and 2 in Arm A Versus Arm C
Description: OS at 1- and 2-year landmark timepoints in Teff-high WT population and ITT-WT population.
Time Frame: Baseline to 2 years or death, whichever occurs first.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 222 | 197
Percentage
  1-Year Teff-high WT Population: number analyzed (Participants) | 110 | 72
  1-Year Teff-high WT Population | 67.48 [60.29 to 74.68] | 56.92 [48.32 to 65.53]
  2-Year Teff-high WT Population: number analyzed (Participants) | 75 | 49
  2-Year Teff-high WT Population | 46.01 [38.36 to 53.66] | 38.74 [30.26 to 47.22]
  1-Year ITT-WT Population | 64.06 [59.02 to 69.11] | 59.89 [54.61 to 65.17]
  2-Year ITT-WT Population: number analyzed (Participants) | 143 | 104
  2-Year ITT-WT Population | 41.45 [36.26 to 46.64] | 31.79 [26.75 to 36.82]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 1-Year ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.2624, Z-test; Difference in Event Free Rate = 4.18, 95% CI 2-sided [-3.13 to 11.48]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 2-Year ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.0088, Z-test; Difference in Event Free Rate = 9.67, 95% CI 2-sided [2.43 to 16.90]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 1-Year Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.0649, Z-test; Difference in Event Free Rate = 10.56, 95% CI 2-sided [-0.65 to 21.77]
Statistical Analysis 4: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); 2-Year Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.2120, Z-test; Difference in Event Free Rate = 7.27, 95% CI 2-sided [-4.15 to 18.69]

17. Secondary Outcome: Time to Deterioration (TTD) in Patient-Reported Lung Cancer Symptoms Determined by European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire-Core 30 (QLQ-C30) Score
Description: EORTC QLQ-C30 is a validated & reliable self-report measure (Aaronson et al.1993;Fitzsimmons et al.1999) that consists of 30 questions that assess 5 aspects of patient functioning (physical,emotional,role, cognitive,and social), 3 symptom scales (fatigue,nausea & vomiting, pain),global health/quality of life,and six single items (dyspnea,insomnia, appetite loss,constipation,diarrhea, and financial difficulties). EORTC QLQ-C30 is scored according to the EORTC scoring manual (Fayers et al. 2001). All EORTC scales and single-item measures are linearly transformed so that each score has a range of 0-100. A high score for a functional/global health status scale represents a high or healthy level of functioning/HRQoL (Health-Related Quality of Life);however a high score for a symptom scale or item represents a high level of symptomatology or problems. A ≥10-point change in the symptoms subscale score is perceived by patients as clinically significant (Osoba et al.1998).
Time Frame: Baseline up to approximately 29 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 348 | 356 | 336
Months
  Dyspnea in Teff-high WT Population: number analyzed (Participants) | 161 | 155 | 129
  Dyspnea in Teff-high WT Population | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Dyspnea in ITT-WT Population | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.6899, Log Rank; Hazard Ratio (HR) = 0.909, 95% CI 2-sided [0.571 to 1.450]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.1043, Log Rank; Hazard Ratio (HR) = 0.671, 95% CI 2-sided [0.413 to 1.089]
Statistical Analysis 3: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT WT; Test type: Superiority — Stratified Analysis; p = 0.1730, Log Rank; Hazard Ratio (HR) = 1.232, 95% CI [0.912 to 1.665]
Statistical Analysis 4: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); ITT WT; Test type: Superiority — Stratified Analysis; p = 0.6145, Log Rank; Hazard Ratio (HR) = 1.084, 95% CI 2-sided [0.792 to 1.483]

18. Secondary Outcome: TTD in Patient-Reported Lung Cancer Symptoms as Determined by EORTC Quality-of-Life Questionnaire-Core Lung Cancer Module 13 (QLQ-LC13) Score
Description: QLQ-LC13 Quality-of-Life Questionnaire Lung Cancer Module incorporates one multiple-item scale to assess dyspnea and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. The EORTC QLQ-LC13 is scored according to the EORTC scoring manual (Fayers et al. 2001). All EORTC scales and single-item measures are linearly transformed so that each score has a range of 0-100. A high score for a functional/global health status scale represents a high or healthy level of functioning/HRQoL (Health-Related Quality of Life); however, a high score for a symptom scale or item represents a high level of symptomatology or problems. A ≥10-point change in the symptoms subscale score is perceived by patients as clinically significant (Osoba et al. 1998).
Time Frame: Baseline up to approximately 29 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 348 | 356 | 336
Months
  Cough in Teff-high WT Population: number analyzed (Participants) | 161 | 155 | 129
  Cough in Teff-high WT Population | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [21.0 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Dyspnea in Teff-high WT Population: number analyzed (Participants) | 161 | 155 | 129
  Dyspnea in Teff-high WT Population | NA [5.6 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [6.3 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Chest Pain in Teff-high WT Population: number analyzed (Participants) | 161 | 155 | 129
  Chest Pain in Teff-high WT Population | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 22.2 [22.2 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 18.4 [18.4 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Arm and/or Shoulder Pain in Teff-high WT: number analyzed (Participants) | 161 | 155 | 129
  Arm and/or Shoulder Pain in Teff-high WT | NA [18.3 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 19.5 [12.5 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [12.7 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Cough in ITT-WT Population | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [21.0 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Dyspnea in ITT-WT Population | 21.9 [9.7 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [10.0 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Arm and/or Shoulder Pain in ITT-WT | NA [18.3 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 19.5 [15.2 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
  Pain in Chest in ITT-WT Population | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. Median is not reached and the confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [22.2 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [18.4 to NA] — Value is not available due to an insufficient number of participants with the event. Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.
Statistical Analysis 1: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Cough for Teff-high WT ITT population; Test type: Superiority — Stratified Analysis; p = 0.8816, Log Rank; Hazard Ratio (HR) = 1.041, 95% CI 2-sided [0.614 to 1.763]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Cough for Teff-high WT ITT Population; Test type: Superiority — Stratified Analysis; p = 0.2995, Log Rank; Hazard Ratio (HR) = 0.741, 95% CI 2-sided [0.419 to 1.309]
Statistical Analysis 3: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Dyspnea in Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.7578, Log Rank; Hazard Ratio (HR) = 0.936, 95% CI 2-sided [0.616 to 1.422]
Statistical Analysis 4: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Dyspnea in Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.8470, Log Rank; Hazard Ratio (HR) = 1.041, 95% CI 2-sided [0.694 to 1.560]
Statistical Analysis 5: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Pain in Chest in Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.1289, Log Rank; Hazard Ratio (HR) = 0.659, 95% CI 2-sided [0.383 to 1.133]
Statistical Analysis 6: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Pain in Chest in Teff-high WT Population; Test type: Superiority — Stratified Analysis; p = 0.2381, Log Rank; Hazard Ratio (HR) = 0.729, 95% CI 2-sided [0.430 to 1.235]
Statistical Analysis 7: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Arm and/or Shoulder Pain in Teff-high WT; Test type: Superiority — Stratified Analysis; p = 0.7163, Log Rank; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.685 to 1.732]
Statistical Analysis 8: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Arm and/or Shoulder Pain in Teff-high WT; Test type: Superiority — Stratified Analysis; p = 0.1502, Log Rank; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.420 to 1.145]
Statistical Analysis 9: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Cough in ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.9568, Log Rank; Hazard Ratio (HR) = 1.010, 95% CI 2-sided [0.713 to 1.430]
Statistical Analysis 10: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Cough in ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.5377, Log Rank; Hazard Ratio (HR) = 0.891, 95% CI 2-sided [0.619 to 1.284]
Statistical Analysis 11: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Dyspnea in ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.4012, Log Rank; Hazard Ratio (HR) = 0.893, 95% CI 2-sided [0.685 to 1.163]
Statistical Analysis 12: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Dyspnea in ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.7149, Log Rank; Hazard Ratio (HR) = 1.050, 95% CI 2-sided [0.809 to 1.363]
Statistical Analysis 13: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Arm and/or Shoulder Pain in ITT-WT; Test type: Superiority — Stratified Analysis; p = 0.7126, Log Rank; Hazard Ratio (HR) = 1.057, 95% CI 2-sided [0.786 to 1.422]
Statistical Analysis 14: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Arm and/or Shoulder Pain in ITT-WT; Test type: Superiority — Stratified Analysis; p = 0.6053, Log Rank; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.675 to 1.258]
Statistical Analysis 15: Comparison: Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Pain in Chest in ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.3134, Log Rank; Hazard Ratio (HR) = 0.829, 95% CI 2-sided [0.576 to 1.194]
Statistical Analysis 16: Comparison: Arm A (Atezolizumab+Paclitaxel+Carboplatin) vs Arm C (Bevacizumab+Paclitaxel+Carboplatin); Pain in Chest in ITT-WT Population; Test type: Superiority — Stratified Analysis; p = 0.6115, Log Rank; Hazard Ratio (HR) = 0.910, 95% CI 2-sided [0.633 to 1.309]

19. Secondary Outcome: Change From Baseline in Patient-Reported Lung Cancer Symptoms Score Using the Symptoms in Lung Cancer (SILC) Scale
Description: The SILC (Symptoms in Lung Cancer) scale was used to assess patient-reported severity of lung cancer symptoms (chest pain, dyspnea, and cough). The SILC scale is a 9-item content validated self-report measure of lung cancer symptoms. It measures severity of cough, dyspnea, and chest pain with a symptom severity score. The SILC questionnaire comprises three individual symptoms (dyspnea, cough, chest pain) and are scored at the individual symptom level, thus have a dyspnea score, chest pain score, and cough score. Each individual symptom score is calculated as the average of responses for the symptom items [e.g. Chest Pain Score=mean (item 1; item 2)]. An increase in score is suggestive of a worsening in symptomology (i.e. frequency or severity). A score change of ≥0.3 points for the dyspnea and cough symptom scores is considered to be clinically significant; whereas a score change of ≥0.5 points for the chest pain score is considered to be clinically significant.
Time Frame: Baseline up to approximately 29 months
Population: No participants were analyzed due to psychometric properties within the NSCLC population are still being determined. Due to quality issues data not analyzed.
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with at least one adverse event.
Time Frame: Baseline up to data cutoff date 7 December 2020 (up to approximately 68 months)
Population: Safety population included all treated patients, defined as randomized patients who received any amount of any component of study treatment.
Measure: Number; unit: Percentage
Arm/Group | Arm C (Bevacizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm A (Atezolizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 394 | 393 | 400
Percentage | 99.0 | 98.2 | 97.8

21. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Time Frame: Baseline up to approximately 29 months
Population: The baseline ADA-evaluable population for each study treatment included patients who had a baseline ADA result. The post-baseline ADA-evaluable population for each study treatment included patients who had at least one post-baseline ADA result and had received at least on dose of that study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin)
Number analyzed (Participants) | 389 | 376
Percentage of Participants | 4.6 | 2.9

22. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Atezolizumab in Arm A and Arm B
Description: The predose samples will be collected on the same day of treatment administration. The infusion duration of atezolizumab will be of 30-60 minutes.
Time Frame: Day 1 of Cycle 1 and 3 (Cycle length=21 days)
Population: The pharmacokinetic-evaluable population is defined as all patients who received any dose of atezolizumab, bevacizumab, carboplatin, or paclitaxel and who had evaluable PK samples post-dose.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin)
Number analyzed (Participants) | 378 | 364
mcg/mL
  Cycle 1 Day 1 | 410 (157) | 414 (127)
  Cycle 3 Day 1: number analyzed (Participants) | 310 | 302
  Cycle 3 Day 1 | 498 (160) | 540 (198)

23. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Atezolizumab Prior to Infusion in Arm A and Arm B
Time Frame: Day 21 of Cycles 1, 2 3, and 7 (Cycle length=21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin)
Number analyzed (Participants) | 354 | 345
mcg/mL
  Cycle 1 Day 21 | 76.4 (37.7) | 80.8 (41.4)
  Cycle 2 Day 21: number analyzed (Participants) | 322 | 319
  Cycle 2 Day 21 | 119 (55.7) | 130 (57.1)
  Cycle 3 Day 21: number analyzed (Participants) | 312 | 307
  Cycle 3 Day 21 | 146 (58.9) | 160 (102)
  Cycle 7 Day 21: number analyzed (Participants) | 230 | 249
  Cycle 7 Day 21 | 219 (89.6) | 220 (99.0)

24. Secondary Outcome: Plasma Concentrations for Carboplatin in Arm A, Arm B, and Arm C
Time Frame: Predose (same day of treatment administration), 5-10 minutes before end of carboplatin infusion, 1 h after carboplatin infusion (infusion duration=15 to 30 minutes) on D1 of Cy1,3 (Cycle length=21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 28 | 35 | 24
ng/mL
  Cy1D1 Pre-dose | NA (NA) — Predose of Cycle 1 Day 1 administration of Carboplatin. | NA (NA) — Predose of Cycle 1 Day 1 administration of Carboplatin. | NA (NA) — Predose of Cycle 1 Day 1 administration of Carboplatin.
  Cy1D1 Before End of Infusion: number analyzed (Participants) | 26 | 32 | 24
  Cy1D1 Before End of Infusion | 18300 (9610) | 18300 (11900) | 17200 (9860)
  Cy1D1 After Infusion: number analyzed (Participants) | 26 | 31 | 22
  Cy1D1 After Infusion | 11700 (5570) | 13900 (14300) | 10100 (5320)
  Cy2D21: number analyzed (Participants) | 19 | 27 | 17
  Cy2D21 | 176 (82.9) | 190 (113) | 143 (73.0)
  Cy3D1 Before End of Infusion: number analyzed (Participants) | 18 | 28 | 16
  Cy3D1 Before End of Infusion | 20900 (8330) | 18700 (9410) | 20600 (12900)
  Cy3D1 After Infusion: number analyzed (Participants) | 20 | 27 | 17
  Cy3D1 After Infusion | 11700 (6990) | 12200 (7480) | 10400 (4150)

25. Secondary Outcome: Plasma Concentrations for Paclitaxel in Arm A, Arm B, and Arm C
Time Frame: Predose (same day of treatment administration), 5-10 minutes before end of paclitaxel infusion, 1 h after paclitaxel infusion (infusion duration=3 h) on D1 of Cy1,3 (Cycle length=21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Atezolizumab+Paclitaxel+Carboplatin) | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 28 | 35 | 24
ng/mL
  Cy1D1 Pre-dose | NA (NA) — Predose of Cycle 1 Day 1 administration of Paclitaxel. | NA (NA) — Predose of Cycle 1 Day 1 administration of Paclitaxel. | NA (NA) — Predose of Cycle 1 Day 1 administration of Paclitaxel.
  Cy1D1 Before End of Infusion: number analyzed (Participants) | 26 | 34 | 24
  Cy1D1 Before End of Infusion | 4850 (2800) | 6440 (3640) | 5560 (2590)
  Cy1D1 After Infusion: number analyzed (Participants) | 27 | 32 | 23
  Cy1D1 After Infusion | 2300 (2790) | 2490 (3020) | 1980 (1780)
  Cy2D21: number analyzed (Participants) | 2 | 3 | 0
  Cy2D21 | NA (NA) — Mean or SD is not reported because more than half of the samples at the specified timepoint are below the limit of quantification. | NA (NA) — Mean or SD is not reported because more than half of the samples at the specified timepoint are below the limit of quantification. |
  Cy3D1 Before End Of Infusion: number analyzed (Participants) | 19 | 25 | 16
  Cy3D1 Before End Of Infusion | 5810 (3610) | 7810 (4510) | 7810 (5160)
  Cy3D1 After Infusion: number analyzed (Participants) | 19 | 27 | 17
  Cy3D1 After Infusion | 1800 (1660) | 2990 (5830) | 1930 (1380)

26. Secondary Outcome: Cmax of Bevacizumab in Arm B and Arm C
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1 (Cycle length=21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 205 | 215
mcg/mL
  Cycle 1 Day 1 | 329 (129) | 323 (95.0)
  Cycle 3 Day 1: number analyzed (Participants) | 154 | 168
  Cycle 3 Day 1 | 413 (126) | 430 (123)

27. Secondary Outcome: Cmin of Bevacizumab in Arm B and Arm C
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 21 (Cycle length=21 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm B (Atezolizumab+Bevacizumab+Paclitaxel + Carboplatin) | Arm C (Bevacizumab+Paclitaxel+Carboplatin)
Number analyzed (Participants) | 325 | 348
mcg/mL
  Cycle 1 Day 1 | NA (NA) — Predose of Cycle 1 Day 1 administration of Bevacizumab. | NA (NA) — Predose of Cycle 1 Day 1 administration of Bevacizumab.
  Cycle 2 Day 21: number analyzed (Participants) | 280 | 316
  Cycle 2 Day 21 | 98.0 (50.9) | 90.4 (36.8)

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date 7 December 2020 (up to approximately 68 months)
Description: The safety population included all treated participants, defined as randomized participants who received any amount of any component of study treatment.
Groups:
- Arm C (Bev+CP): Bevacizumab+Paclitaxel+Carboplatin
- Arm B (Atezo+Bev+CP): Atezolizumab+Bevacizumab+Paclitaxel+Carboplatin
- Arm A (Atezo+CP): Atezolizumab+Paclitaxel+Carboplatin
Arm/Group | Arm C (Bev+CP) | Arm B (Atezo+Bev+CP) | Arm A (Atezo+CP)
All-Cause Mortality (participants affected / at risk) | 311/394 | 285/393 | 293/400
Serious Adverse Events (participants affected / at risk) | 142/394 | 190/393 | 170/400
Other Adverse Events (participants affected / at risk) | 381/394 | 375/393 | 385/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Bev+CP) (N=394) | Arm B (Atezo+Bev+CP) (N=393) | Arm A (Atezo+CP) (N=400)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 5 (6)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 17 (18) | 27 (30) | 13 (13)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1)
NORMOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
AUTOIMMUNE MYOCARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (3) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 2 (2) | 1 (1)
ADRENOCORTICAL INSUFFICIENCY ACUTE (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
DIABETES INSIPIDUS (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOPHYSITIS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
SECONDARY ADRENOCORTICAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 10 (11) | 8 (8)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
FAECALOMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
GLOSSODYNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL ANGINA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
INTESTINAL INFARCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 7 (7) | 1 (1)
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 5 (5) | 4 (5)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
CATHETER SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 6 (7) | 4 (4) | 1 (2)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 2 (2) | 2 (2) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2) | 2 (2) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 1 (1)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 8 (8) | 6 (6)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (2) | 2 (2)
HYPERSENSITIVITY (Immune system disorders) | 2 (2) | 1 (2) | 1 (1)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BONE ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
BURSITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTERITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGIC PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS A (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
INFECTED SKIN ULCER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
KLEBSIELLA SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PAROTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 18 (19) | 28 (30) | 21 (23)
PNEUMONIA ADENOVIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
PROSTATIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYOPNEUMOTHORAX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
RESPIRATORY TRACT INFECTION FUNGAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SCROTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 5 (5) | 3 (4) | 3 (3)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 4 (4)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 2 (2) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 7 (9) | 3 (3)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MARROW HYPERPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
TUMOUR PSEUDOPROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 5 (5) | 2 (2)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
FOCAL DYSCOGNITIVE SEIZURES (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 5 (5) | 2 (3)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DELUSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 3 (3) | 2 (2)
GLOMERULONEPHROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
PRERENAL FAILURE (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
RENAL INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
BRONCHOSTENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 3 (4)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
IMMUNE-MEDIATED PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 8 (8)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 4 (4)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5) | 8 (8)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
PULMONARY NECROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
VERTEBROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ANEURYSM (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
DIABETIC VASCULAR DISORDER (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
EMBOLISM VENOUS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Bev+CP) (N=394) | Arm B (Atezo+Bev+CP) (N=393) | Arm A (Atezo+CP) (N=400)
ANAEMIA (Blood and lymphatic system disorders) | 104 (124) | 116 (134) | 146 (183)
LEUKOPENIA (Blood and lymphatic system disorders) | 14 (17) | 14 (20) | 20 (35)
NEUTROPENIA (Blood and lymphatic system disorders) | 70 (107) | 72 (111) | 60 (85)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 45 (64) | 53 (74) | 49 (78)
HYPOTHYROIDISM (Endocrine disorders) | 13 (13) | 50 (56) | 33 (40)
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 (24) | 36 (48) | 29 (36)
CONSTIPATION (Gastrointestinal disorders) | 92 (115) | 122 (151) | 103 (128)
DIARRHOEA (Gastrointestinal disorders) | 98 (133) | 125 (221) | 82 (137)
DRY MOUTH (Gastrointestinal disorders) | 6 (6) | 20 (22) | 13 (16)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 9 (11) | 20 (20) | 11 (13)
NAUSEA (Gastrointestinal disorders) | 124 (177) | 149 (223) | 130 (210)
STOMATITIS (Gastrointestinal disorders) | 24 (30) | 54 (73) | 23 (27)
VOMITING (Gastrointestinal disorders) | 67 (105) | 71 (99) | 69 (92)
ASTHENIA (General disorders) | 80 (107) | 84 (143) | 76 (127)
CHEST PAIN (General disorders) | 28 (32) | 35 (37) | 38 (44)
FATIGUE (General disorders) | 107 (125) | 137 (157) | 111 (129)
MALAISE (General disorders) | 11 (13) | 27 (43) | 20 (27)
MUCOSAL INFLAMMATION (General disorders) | 24 (27) | 38 (42) | 10 (10)
OEDEMA PERIPHERAL (General disorders) | 19 (20) | 35 (42) | 29 (33)
PAIN (General disorders) | 17 (17) | 26 (31) | 22 (23)
PYREXIA (General disorders) | 34 (44) | 67 (88) | 53 (66)
BRONCHITIS (Infections and infestations) | 16 (17) | 28 (37) | 15 (16)
NASOPHARYNGITIS (Infections and infestations) | 17 (18) | 27 (34) | 31 (50)
PNEUMONIA (Infections and infestations) | 15 (17) | 19 (22) | 21 (23)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 (20) | 37 (56) | 24 (43)
URINARY TRACT INFECTION (Infections and infestations) | 28 (37) | 35 (57) | 37 (51)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 20 (24) | 30 (45) | 22 (26)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 18 (19) | 30 (48) | 22 (29)
NEUTROPHIL COUNT DECREASED (Investigations) | 34 (72) | 49 (87) | 33 (64)
PLATELET COUNT DECREASED (Investigations) | 44 (76) | 57 (84) | 41 (59)
WEIGHT DECREASED (Investigations) | 42 (46) | 52 (56) | 29 (32)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 20 (39) | 26 (42) | 17 (27)
DECREASED APPETITE (Metabolism and nutrition disorders) | 86 (102) | 119 (157) | 100 (129)
DEHYDRATION (Metabolism and nutrition disorders) | 15 (16) | 33 (42) | 7 (7)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 16 (18) | 36 (47) | 24 (30)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 25 (29) | 55 (76) | 38 (49)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 17 (20) | 23 (32) | 13 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 102 (155) | 130 (227) | 105 (175)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 43 (50) | 57 (67) | 51 (70)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 19 (19) | 23 (33) | 16 (18)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 (8) | 20 (24) | 10 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 53 (81) | 69 (118) | 67 (104)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 32 (43) | 50 (63) | 45 (52)
DIZZINESS (Nervous system disorders) | 26 (31) | 27 (34) | 28 (39)
DYSGEUSIA (Nervous system disorders) | 19 (24) | 24 (27) | 15 (16)
HEADACHE (Nervous system disorders) | 53 (65) | 70 (87) | 41 (49)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 67 (77) | 92 (105) | 104 (117)
PARAESTHESIA (Nervous system disorders) | 44 (50) | 53 (59) | 37 (42)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 54 (59) | 65 (73) | 58 (65)
ANXIETY (Psychiatric disorders) | 22 (23) | 31 (31) | 23 (23)
DEPRESSION (Psychiatric disorders) | 13 (13) | 25 (26) | 15 (16)
INSOMNIA (Psychiatric disorders) | 38 (41) | 42 (43) | 50 (56)
PROTEINURIA (Renal and urinary disorders) | 63 (81) | 80 (128) | 9 (13)
COUGH (Respiratory, thoracic and mediastinal disorders) | 77 (94) | 86 (107) | 82 (99)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 27 (27) | 11 (12)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 60 (66) | 67 (81) | 86 (107)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 86 (108) | 67 (89) | 17 (22)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 21 (24) | 16 (27)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 22 (25) | 9 (10)
ALOPECIA (Skin and subcutaneous tissue disorders) | 180 (183) | 188 (195) | 180 (182)
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 (9) | 29 (31) | 24 (28)
PRURITUS (Skin and subcutaneous tissue disorders) | 25 (29) | 58 (76) | 52 (72)
RASH (Skin and subcutaneous tissue disorders) | 28 (34) | 72 (92) | 71 (94)
HYPERTENSION (Vascular disorders) | 87 (102) | 104 (149) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT02366143/Prot_001.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT02366143/SAP_000.pdf